CLINICAL TRIAL: NCT02689401
Title: MRI Iron Oxide Imaging for Lymph Node Staging in Esophageal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Awaiting additional safety data
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Yolonda L. Colson, MD, PhD, Yolonda Colson MD PhD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-419
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; lymph nodes tumor
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ferumoxtyol (Feraheme) with MRI (Experimental): Patients will undergo a pre-contrast MRI followed by a pre determined dose of of IV Ferumoxyto. Post-contrast MRI imaging will be performed immediately following Ferumoxytol infusion and 48 hours after Ferumoxytol administration with subsequent image analysis.
  Interventions: Drug: Ferumoxytol; Device: MRI 3T scanner

INTERVENTIONS:
Drug: Ferumoxytol
  Other Names: Feraheme
Device: MRI 3T scanner

SUMMARY:
This research study is evaluating a new imaging method using MRI (magnetic resonance imaging) to evaluate lymph nodes for evidence of tumor spread from esophageal cancer. This MRI study involves an intravenous contrast called Ferumoxytol (FerahemeTM).

DETAILED DESCRIPTION:
This research study is a Pilot clinical trial, which is the first time investigators are examining this study intervention.

This study tests the safety of the investigational intervention (MRI imaging with Ferumoxytol) and assesses the feasibility of identifying malignant lymph nodes (lymph nodes that have tumor in them) by comparing the experimental MRI findings with the final pathology report from surgery.

This iron-based agent currently has approval from the U.S. Food and Drug Administration (FDA) for use in iron replacement therapy, however, its use in MRI imaging is not FDA-approved and is thus experimental in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants may have histologically confirmed esophageal cancer or lesion suspicious for esophageal cancer which is deemed surgically resectable.
* Patients eligible for the trial may have previously completed neoadjuvant chemoradiation per standard protocols prior to MRI imaging, without any limitations on dose, duration or type of prior treatment as this is not the focus of the current study.
* Eligible patients must be 18 years or older in order to consent for this trial. Individuals under the age of 18 are excluded because safety studies including dosing or adverse event data in this population are currently not available.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with known allergies or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharides
* Individuals who are pregnant or lactating. As part of their routine preoperative testing, all women of child bearing age receive a pregnancy test. The research staff will follow up on these results in order to determine eligibility. Women who have had a hysterectomy or have not had menses for > 24 months will not be required to undergo a pregnancy test. Pregnant women are excluded from this study because there is unknown risk associated with Ferumoxytol (US FDA Risk Category C: there are no controlled studies in women, or no studies are available in either animals or women). Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding women will be excluded from this study
* Iron saturation above the upper limit of normal
* Individuals with known clinical conditions that may lead to iron overload including hemochromatosis, cirrhosis, or sickle cell disease
* Individuals with a contraindication to MRI, such as the presence of metallic prostheses or implanted metal device (e.g. infusion pump, defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of using MRI-ferumoxytol for the identification of metastatic lymph nodes in patients with esophageal cancer | 2 years
  Feasibility is determined by the ability of the radiologist to identify esophageal associated lymph nodes and which ones may be metastatic based on the uptake of ferumoxytol. Positive nodes are identified by the radiologist based on altered signal in those with ferumoxytol uptake compared to the signal normal lymph nodes on MRI
Assess the safety of intravenous ferumoxytol for the use in esophageal cancer patients | 2 years
  Safety is determined by none of the 10 patients developing a grade 3 or 4 reaction as per the Common Toxicity Criteria scale (NCI-CTCAE version 4.0)

SECONDARY OUTCOMES:
Determine the accuracy of MRI-ferumoxytol for the identification of positive metastatic nodes in patients with esophageal cancer | 2 years
  Accuracy is determined by the positive metastatic nodes identified on MRI as compared to those found on pathologic examination

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda Colson, MD PhD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No